CLINICAL TRIAL: NCT02203539
Title: The Influence of Different Light Exposures on Endurance Performance, Handgrip Strength and Reaction Time in Consideration of the Chronotype.
Brief Title: The Influence of Light Exposure on Exercise Performance Dependent on Chronotype.
Acronym: EX-Light
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Arno Schmidt-Trucksäss, Prof Arno Schmidt-Trucksäss, MD, MA, University of Basel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EKNZ 2014-056
Record Dates: First submitted 2014-04-16; First posted 2014-07-30 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Endurance Performance; Reaction Time; Muscle Strength
Keywords: circadian rhythm; light exposure; exercise capacity; endurance; strength; reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- bright light (Experimental): Intervention: exposure to bright light
  Interventions: Other: exposure to bright light
- blue-enriched light (Experimental): Intervention: exposure to blue-enriched light
  Interventions: Other: exposure to blue-enriched light
- normal light (Experimental): Intervention: exposure to normal light
  Interventions: Other: exposure to normal light

INTERVENTIONS:
Other: exposure to normal light — exposure for 60 minutes in duration
  Arms: normal light
Other: exposure to bright light — exposure to bright light for 60 minutes of duration
  Arms: bright light
Other: exposure to blue-enriched light — exposure to blue-enriched light for 60 minutes of duration
  Arms: blue-enriched light

SUMMARY:
The purpose of this study is to determine if an exposure to light in the evening has a positive influence on physical performance regarding endurance, strength and reaction time.

ELIGIBILITY:
Inclusion criteria:

* BMI 18 to 30 kg/m2
* endurance performance >= 55 ml/min/kg peak oxygen uptake

Exclusion criteria:

* cardiovascular disease
* renal dysfunction
* shiftworking
* travels over time zones in the last 4 weeks
* high blood pressure (systolic blood pressure >170mmHg, diastolic blood pressure >100mmHg)
* depression

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Work performed in kilo Joule (kJ) during the time trial ergometer test adjusted for the VO2peak. | The outcome measure will be assesed at the end of the 12minute time trial ergometer test.
  Participants will perform one baseline test (ergometer ramp test) and seven days later a twelve minute lasting ergometer time trial test which starts 10 minutes after an exposure to light for 60minutes. The work performed in kilo Joule during the time trial ergometer test will be assesed at the end of the time trial and will be the main outcome measure and adjusted for the VO2peak meausred during the baseline test.

SECONDARY OUTCOMES:
Reaction time in milliseconds (ms) | Reaction time task will be performed at baseline (20 to 15 minutes before the light exposure) and 0 to minutes after the light exposure which will be the secondary outcome measure.
  Participants will perform one baseline reaction time task 20 to 15 minutes before the light exposure. 0 to 5 minutes after the 60 minutes lasting light exposure they will perform the reaction task again. The time in milliseconds from the reaction task after the light exposure will be the secondary outcome measure and adjusted for the baseline test before light exposure.
Maximum handgrip strength in kilo gramm (kg) | Maximum handgrip strength will be tested at baseline (15 to 10 minutes before the light exposure) and 5 to 10 minutes after the 60 minutes lasting light exposure.
  Participants will perform one baseline maximum hand grip strength test 15 to 10 minutes before the 60 minutes lasting light exposusre and perform a second test, which will be the outcome measure 5 to 10 minutes after the light exposure. The strength in kg will be adjusted for the strength in kg measured at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Arno Schmidt-Trucksäss, Prof Dr, Principal Investigator — Departement of Sports, Exercise and Health, University of Basel
Locations (1):
- Department for Sport, Exercise and Health, Section Sports and Exercise Medicine, University of Basel, Basel, Switzerland